CLINICAL TRIAL: NCT07311174
Title: Can Psychodrama Improve Aggressive Behavior and Social Adjustment? A Randomized Controlled Trial Among Male Adolescents in a Tropical Developing Region
Brief Title: Can Psychodrama Improve Aggressive Behavior and Social Adaptation in Adolescent Boys?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerman University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Parvin Rezaei-Gazki, faculty member, Kerman University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IR.IAU.BA.REC.1402.049
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Aggressive Behavior
MeSH Terms: conditions — Aggression | interventions — Psychodrama

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodrama (Experimental): Participants received a 10-session structured psychodrama intervention based on Blatner's protocol. Sessions were held weekly for 90 minutes.
  Interventions: Behavioral: Psychodrama
- Standard school program (Active Comparator): Participants continued with their standard school educational program. They received no additional sessions, therapy, or intervention during the 10-week study period.
  Other: Standard Care
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Psychodrama — Participants received a 10-session structured psychodrama intervention based on Blatner's protocol. Sessions were held weekly for 90 minutes.
  Arms: Psychodrama
Other: Control — The control group recieved no intervention during 10 weeks.
  Arms: Standard school program

SUMMARY:
This randomized controlled trial evaluated the effectiveness of a 10-session psychodrama intervention on reducing aggressive behavior and improving social adjustment among male adolescents with high aggression and low social adjustment in Bandar Abbas, southern Iran. Twenty-two eligible students were randomly assigned to either a psychodrama intervention group or a comparison group. Outcomes were assessed using the Buss-Perry Aggression Questionnaire and the Bell Adjustment Inventory before and after the intervention.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted in 2023 among male adolescents aged 11-15 years at a public secondary school in Bandar Abbas, a tropical hot desert region in southern Iran. Students were screened using the Buss-Perry Aggression Questionnaire (BPAQ) and the Bell Adjustment Inventory (BAI). Those with high aggression (BPAQ >117) and low social adjustment (BAI score 16-20) were eligible.

Twenty-two students meeting eligibility criteria were randomly assigned in a 1:1 ratio to either the psychodrama intervention group (n=11) or the comparison group (n=11). One participant in the intervention group dropped out, resulting in final analysis of 21 participants.

The intervention consisted of 10 weekly 90-minute psychodrama sessions based on Blatner's protocol, including role-playing, mirroring, soliloquy, storytelling, future projection, and relaxation exercises. The comparison group received no intervention during the study period but was offered the program after study completion.

Primary outcomes were aggression (measured by BPAQ) and social adjustment (measured by BAI), assessed at baseline and post-intervention. Data were analyzed using ANCOVA and repeated measures ANOVA.

ELIGIBILITY:
Inclusion criteria:

* Male, 7th or 8th-grade student (aged 11-13).
* BPAQ score > 117.
* BAI score between 16 and 20.
* Able to commute to after-school classes.
* Parental informed consent obtained.

Exclusion criteria:

* Physical disability or severe illness.
* History of major psychiatric disorders or current psychiatric medication use.
* Unwillingness to participate or missing >2 sessions.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Bell Adjustment Inventory | Pre-intervention and immediately post-intervention (10 weeks)
  Higher scores= Worst outcome (Poorer adjustment).
Buss-Perry Aggression Questionnaire | Pre-intervention and immediately post-intervention (10 weeks)
  Higher scores= Worst outcome (Greater aggression).

CONTACTS AND LOCATIONS:
Locations (1):
- Kerman University of Medical Sciences, Kerman, Iran

IPD SHARING:
Plan to Share IPD: Undecided